CLINICAL TRIAL: NCT02284802
Title: Early Detection of Tumors of the Digestive Tract by Confocal Endomicroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fauze Maluf Filho (Other)
Responsible Party: Sponsor-Investigator, Fauze Maluf Filho, MD, PHD, Instituto do Cancer do Estado de São Paulo
Organization: Instituto do Cancer do Estado de São Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NP354/13
Record Dates: First submitted 2014-11-02; First posted 2014-11-06 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Barrett Esophagus; Gastric Antrectomy Partial; Biliary Duct Stricture; Pancreatic Duct Stricture; Colorectal Polyps; Esophageal Neoplasms; Head and Neck Neoplasms
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Confocal endomicroscopy (Experimental): Pts will be submitted to confocal endomicroscopy examination of the area of interest during endoscopy. A presumptive diagnosis will be made. This diagnosis will be compared to the definitive histologic diagnosis provided by endoscopic biopsies of the area of interest.
  Interventions: Procedure: Confocal endomicroscopy

INTERVENTIONS:
Procedure: Confocal endomicroscopy — Confocal endomicroscopy examination during endoscopy

SUMMARY:
Confocal endomicroscopy is an emerging technique that allows in vivo imaging of cells and tissue structures of the gastrointestinal mucosa, with a magnification of about 1000 times, guiding optical biopsies in real time. Confocal endomicroscopy represents technique that combines conventional white light image with the confocal microscope probe, thereby allowing examination of the surface epithelium in vivo and histological diagnosis during endoscopy. Among the applications already established for its use, stand out diagnosis of Barrett's esophagus, gastric atrophy and intestinal metaplasia, celiac disease, differentiation of hyperplastic adenomatous polyps of the colon, microscopic colitis and follow-up of patients with inflammatory disease, reducing the need for endoscopic biopsies. The CLE can still detect molecular changes effectively improving the endoscopic diagnosis. This pilot project consists of 07 subprojects which the technology of confocal endomicroscopia will be evaluated and compared with the histological results of biopsy or surgical specimens:

1. confocal endomicroscopy for the diagnosis of high-grade dysplasia and superficial esophageal adenocarcinoma in patients with Barrett's esophagus 2 Diagnosis of superficial esophageal squamous cell carcinoma in patients with head and neck cancer by confocal endomicroscopy 3 Detect the presence of premalignant lesions in the gastric stump in patients with reflux alkaline gastritis after partial gastrectomy 4. detect lesions in the gastric mucosa of patients with familial history of gastric cancer 5 Biliary Strictures: differential diagnosis by confocal endomicroscopia 6 confocal Endomicroscopy of cystic neoplasms of the pancreas 7 Contribution of confocal endomicroscopy for the differential diagnosis of colorectal polyps The project aims to deploy the structure of the Confocal endomicroscopy Endoscopy ICESP, for performing in vivo histological examinations of the digestive tract, biliary tract and pancreas. All research groups involved in the early detection of tumors of the esophagus, stomach, biliary tract, pancreas, colon and rectum may benefit from the implementation of this methodology.

DETAILED DESCRIPTION:
Confocal Endomicroscopy procedure: eligible patients which consent to participate in the study will be submitted to endoscopic procedures under conscious or deep sedation. The patients will receive an intravenous injection of 2.5-5 mL of 10% sodium fluorescein at the beginning of the endoscopic procedure. The endoscope will target the area of interest and the confocal probe will be passed through the endoscope biopsy channel. The probe will gently and perpendicularly touch the mucosal surface of the area of the interest. The images will be recorded and a presumptive diagnosis will be made. The area of interest will be biopsied and the histology results will be considered the diagnostic gold standard method. We will calculate the diagnostic accuracy of the presumptive diagnosis provided by the confocal endomicroscopy examination.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old
* Clinical conditions for the proposed endoscopic procedure
* Sign the informed consent

Exclusion Criteria:

* History of anaphylactic reactions to fluorescein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
accuracy of confocal endomicroscopy | Less than 7 days
  Diagnostic accuracy of confocal endomicroscopy for the early detection of tumors of the digestive tract

CONTACTS AND LOCATIONS:
Overall Officials: Fauze Maluf-FIlho, MD, PHD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, Brazil

REFERENCES:
- [Result] Safatle-Ribeiro AV, Baba ER, Faraj SF, Rios JT, de Lima MS, Martins BC, Geiger SN, Pennacchi C, Gusman C, Kawaguti FS, Uemura RS, de Melo ES, Ribeiro U Jr, Maluf-Filho F. Diagnostic accuracy of probe-based confocal laser endomicroscopy in Lugol-unstained esophageal superficial lesions of patients with head and neck cancer. Gastrointest Endosc. 2017 Jun;85(6):1195-1207. doi: 10.1016/j.gie.2016.09.031. Epub 2016 Sep 30. PMID 27697445
- [Result] Safatle-Ribeiro AV, Ryoka Baba E, Corsato Scomparin R, Friedrich Faraj S, Simas de Lima M, Lenz L, Costa Martins B, Gusmon C, Shiguehissa Kawaguti F, Pennacchi C, Zilberstein B, Ribeiro U Jr, Maluf-Filho F. Probe-based confocal endomicroscopy is accurate for differentiating gastric lesions in patients in a Western center. Chin J Cancer Res. 2018 Oct;30(5):546-552. doi: 10.21147/j.issn.1000-9604.2018.05.08. PMID 30510366
- [Result] Baba ER, Safatle-Ribeiro AV, Paduani GF, Giovannini M, Maluf-Filho F. Probe-based confocal laser endomicroscopy for the differential diagnosis of gastric tubular adenoma and intestinal metaplasia in a patient with severe atrophic pangastritis. Gastrointest Endosc. 2016 Jul;84(1):183. doi: 10.1016/j.gie.2016.02.033. Epub 2016 Mar 3. No abstract available. PMID 26949002
- [Result] Safatle-Ribeiro AV, Marques CFS, Pires C, Arraes L, Baba ER, Meirelles L, Kawaguti FS, da Costa Martins B, Lenz LT, de Lima MS, Gusmon-Oliveira CC, Ribeiro U Jr, Maluf-Filho F, Nahas SC. Diagnosis of Clinical Complete Response by Probe-Based Confocal Laser Endomicroscopy (pCLE) After Chemoradiation for Advanced Rectal Cancer. J Gastrointest Surg. 2021 Feb;25(2):357-368. doi: 10.1007/s11605-020-04878-y. Epub 2021 Jan 14. PMID 33443686
- [Result] Scomparin RC, Bento LH, Batista CP, Martins BC, Lenz L, Baba ER, Safatle-Ribeiro AV, Maluf-Filho F. Application of confocal endomicroscopy in the diagnostic elucidation of pancreatic cyst. Rev Assoc Med Bras (1992). 2018 Oct;64(10):885-887. doi: 10.1590/1806-9282.64.10.885. No abstract available. PMID 30517234
- [Result] Bastos VR, Safatle-Ribeiro AV, Baba ER, da Costa Martins B, Maluf-Filho F. The impact of probe-based confocal endomicroscopy on the management of indeterminate bile duct strictures. VideoGIE. 2017 Dec 9;3(1):26-27. doi: 10.1016/j.vgie.2017.10.003. eCollection 2018 Jan. No abstract available. PMID 29905177
- [Derived] Safatle-Ribeiro AV, Ribeiro U Jr, Lata J, Baba ER, Lenz L, da Costa Martins B, Kawaguti F, Moura RN, Pennacchi C, Gusmon C, de Lima MS, de Paulo GA, Nahas CS, Marques CF, Imperiale AR, Cotti GC, Maluf-Filho F, Nahas SC. The Role of Probe-Based Confocal Laser Endomicroscopy (pCLE) in the Diagnosis of Sustained Clinical Complete Response Under Watch-and-Wait Strategy After Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Adenocarcinoma: a Score Validation. J Gastrointest Surg. 2023 Sep;27(9):1903-1912. doi: 10.1007/s11605-023-05732-7. Epub 2023 Jun 8. PMID 37291428